CLINICAL TRIAL: NCT01692301
Title: A Randomized, Double-blind 52-week Study to Evaluate the Safety and Efficacy of an LCZ696 Regimen Compared to an Olmesartan Regimen on Arterial Stiffness Through Assessment of Central Blood Pressure in Elderly Patients With Hypertension
Brief Title: Study of the Safety and Efficacy of LCZ696 on Arterial Stiffness in Elderly Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696A2216; 2012-002899-14 (EudraCT Number)
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Hypertension
Keywords: hypertension, elderly, central aortic pulse pressure, central pulse pressure, pulse wave velocity
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; olmesartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LCZ696 (sacubitril/valsartan) (Experimental): Randomized patients received LCZ696 once daily for four weeks, then they force-titrated to a higher dose at Week 4 and stayed on this dose of LCZ696 once daily for the remainder of the treatment period. At week 12, patients with uncontrolled BP allowed to have amlodipine then hydrochlorothiazide (HCTZ) added at intervals of 4 weeks from Week 12 up to Week 24. To maintain the double dummy, double-blind design, 2 tablets (LCZ696, its matching placebo) and 1 capsule (olmesartan matching placebo) were given during the entire study.
  Interventions: Drug: LCZ696; Drug: LCZ696 matching placebo; Drug: Olmesartan matching placebo; Drug: amlodipine; Drug: hydrochlorothiazide
- Olmesartan (Active Comparator): Randomized patients received olmesartan once daily for four weeks, then force-titrated to a higher dose at Week 4 and stayed on this dose of olmesartan once daily for the remainder of the treatment period. At week 12, patients with uncontrolled BP allowed to have amlodipine then hydrochlorothiazide (HCTZ) added at intervals of 4 weeks from Week 12 up to Week 24. To maintain the double dummy, double-blind design, 2 tablets (LCZ696 matching placebo) and 1 capsule (olmesartan) were given during the entire study.
  Interventions: Drug: Olmesartan; Drug: LCZ696 matching placebo; Drug: amlodipine; Drug: hydrochlorothiazide

INTERVENTIONS:
Drug: LCZ696 — 200 mg tablet
  Other Names: sacubitril/valsartan
  Arms: LCZ696 (sacubitril/valsartan)
Drug: Olmesartan — 20 mg and 40 mg capsules
  Arms: Olmesartan
Drug: LCZ696 matching placebo — LCZ696 Matching Placebo tablet
Drug: Olmesartan matching placebo — Olmesartan matching placebo capsule
  Arms: LCZ696 (sacubitril/valsartan)
Drug: amlodipine — amlodipine 2.5 mg or 5 mg tablets
Drug: hydrochlorothiazide — hydrochlorothiazide 6.25mg, 12.5mg, or 25 mg tablets

SUMMARY:
The study examined the efficacy of LCZ696 in comparison to the ARB olmesartan on Central Aortic Systolic Blood Pressure (CASP) and other measures of central hemodynamics and arterial stiffness in elderly patients with an elevated systolic blood pressure (SBP) and widened pulse pressure (PP).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female patients ≥ 60 years of age.
2. Patients with essential hypertension, untreated or currently taking antihypertensive therapy.
3. Untreated patients must have an office msSBP ≥150 mmHg and <180 mmHg at Visit 101 and Visit 201 if they are newly diagnosed or have not been treated with antihypertensive drugs for the 4 weeks prior to Visit 1.
4. Treated patients must have an office msSBP ≥140 mmHg and <180 mmHg at Visit 102 (or Visit 103) and msSBP ≥150 mmHg and <180 mmHg at Visit 201 if they have been treated with antihypertensive drugs for the 4 weeks prior to Visit 1.
5. All patients must have pulse pressure >60 mmHg at Visit 201. Pulse pressure is defined as msSBP- msDBP.
6. Patients must have a difference in msSBP within +/-15 mmHg between Visit 201 (randomization) and the visit immediately prior to Visit 201.

Key Exclusion Criteria:

1. Malignant or severe hypertension (grade 3 of WHO classification; msDBP ≥110 mmHg and/or msSBP ≥ 180 mmHg)
2. History of angioedema, drug-related or otherwise.
3. History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension.
4. Transient ischemic cerebral attack (TIA) during the 12 months prior to Visit 1 or any history of stroke.
5. History of myocardial infarction, coronary bypass surgery or any percutaneous coronary intervention (PCI) during the 12 months prior to Visit 1.
6. History of atrial fibrillation or atrial flutter during the 3 months prior to Visit 1, or active atrial fibrillation or atrial flutter on the ECG at screening.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (41):
- United States (11):
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Pasadena, Texas
- Argentina (3):
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Colombia (2):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla
- Novartis Investigative Site, Paris, France
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Nuremberg
- Greece (2):
  - Novartis Investigative Site, Athens, Athens
  - Novartis Investigative Site, Thessaloniki, Greece
- Italy (3):
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, San Daniele del Friuli, UD
- Novartis Investigative Site, Shimotsuke, Tochigi, Japan
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- South Korea (2):
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
- Spain (8):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Centelles, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Port de Sagunt, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC

REFERENCES:
- [Derived] Williams B, Cockcroft JR, Kario K, Zappe DH, Cardenas P, Hester A, Brunel P, Zhang J. Rationale and study design of the Prospective comparison of Angiotensin Receptor neprilysin inhibitor with Angiotensin receptor blocker MEasuring arterial sTiffness in the eldERly (PARAMETER) study. BMJ Open. 2014 Feb 4;4(2):e004254. doi: 10.1136/bmjopen-2013-004254. PMID 24496699

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Started | 229 ("Started" indicates patients in randomized, full analysis and safety set) | 225
Completed | 184 | 183
Not Completed | 45 | 42
Not completed — Adverse Event | 15 | 12
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 0 | 5
Not completed — Non-compliance with study treatment | 1 | 2
Not completed — Protocol deviation | 9 | 2
Not completed — Patient/guardian decision | 16 | 15
Not completed — Technical problems | 0 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set - All patients who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan | Total
Number analyzed (Participants) | 229 | 225 | 454
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (5.73) | 67.2 (5.97) | 67.7 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 107 | 217
  Male | 119 | 118 | 237

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Central Aortic Systolic Pressure (CASP) at 12 Weeks
Description: Central aortic blood pressure was derived from peripheral pressure waveforms recorded noninvasively from the brachial artery using a cuff-based device. This technique uses the brachial pressure and a signal processing algorithm to transform brachial signals into central blood pressure (BP) waveforms. When the aortic pressure waveform was derived, key pulse wave analysis (PWA) parameters, such as CASP was calculated by the system software.
  At the first study visit, the arm with the highest systolic blood pressure (SBP) was used for all subsequent PWA. Brachial PWA measurements were performed on the same arm that the office blood pressures were taken. Two pulse waveform measurements, meeting all quality control criteria were captured at baseline and at week 12 visits.
Time Frame: baseline, 12 weeks
Population: Full analysis set (FAS): All patients who were randomized. This endpoint included number of patients who had values at both baseline and endpoint (week 12).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 207 | 206
mmHg | -12.57 (1.01) | -8.90 (1.01)
Statistical Analysis 1: Comparison: LCZ696 (Sacubitril/Valsartan) vs Olmesartan; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Net) = -3.66, 95% CI 2-sided [-6.45 to -0.87], Standard Error of Mean 1.42

2. Secondary Outcome: Change From Baseline in Mean Central Pulse (CPP) Pressure
Time Frame: Baseline, 12 weeks, and 52 weeks
Population: Full analysis set (FAS): All patients who were randomized. This endpoint included number of patients who had values at both baseline and endpoint (week 12, week 52). Four patients did not have a successful CASP assessment at Week 12 but passed quality check at Week 52, thus 4 more patients were included in the Week 52 Endpoint analysis
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to Week 12 (n = 207, 206) | -6.41 (0.69) | -3.96 (0.69)
  Baseline to Week 52 (n = 209, 208) | -7.16 (0.69) | -6.65 (0.69)

3. Secondary Outcome: Change From Baseline in Mean Pulse Wave Velocity (PWV)
Description: Pulse wave velocity recordings were performed on patient while in a supine, face-up position.
  Tonometry was performed on the carotid simultaneously with the cuff inflation over the femoral artery. Two pulse wave velocity measures, meeting all quality control criteria were captured at baseline, week 12 and week 52.
Time Frame: baseline, 12 weeks, and 52 weeks
Population: Full analysis set (FAS): All patients who were randomized. This endpoint included number of patients who had values at both baseline and endpoint (week 12 , week 52).
Measure: Least Squares Mean (Standard Error); unit: meter/second
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
meter/second
  Baseline to week 12 (n= 192, 196) | -0.68 (0.12) | -0.57 (0.12)
  Baseline to week 52 ( n= 199, 199) | -0.83 (0.13) | 0.77 (0.13)

4. Secondary Outcome: Change From Baseline in Mean Central Aortic Systolic Pressure (CASP) at 52 Weeks
Description: as for outcome 1
Time Frame: baseline, 52 weeks
Population: Full analysis set (FAS): All patients who were randomized. This endpoint included number of patients who had values at both baseline and endpoint (week 52). Four patients did not have a successful CASP assessment at Week 12 but passed quality check at Week 52, thus 4 more patients were included in the Week 52 Endpoint analysis.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 209 | 208
mmHg | -16.18 (0.96) | -14.70 (0.96)

5. Secondary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP)
Description: At the first study visit, the patient had his/her blood pressure (BP) measured in both arms; the arm in which the highest sitting SBP was found was used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for 5 minutes, SBP were measured 3 times using a standard mercury sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1- to 2-minute intervals and the mean of those 3 measurements was used as the average sitting office BP for that visit.
Time Frame: baseline, 12 weeks, and 52 weeks
Population: Full analysis set (FAS): All patients who were randomized. This endpoint included number of patients who had values at both baseline and endpoints (week 12, week 52).
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n=226, 222) | -20.84 (1.06) | -14.57 (1.07)
  Baseline to week 52 (n=226,223) | -23.91 (0.98) | -21.45 (0.99)

6. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP)
Description: At the first study visit, the patient had his/her blood pressure (BP) measured in both arms; the arm in which the highest sitting SBP was found was used for all subsequent readings throughout the study. At each study visit, after the patient had been sitting for 5 minutes, DBP were measured 3 times using a standard mercury sphygmomanometer and appropriate size cuff. The repeat sitting measurements were made at 1- to 2-minute intervals and the mean of those 3 measurements was used as the average sitting office BP for that visit.
Time Frame: baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n=226, 222) | -7.86 (0.58) | -5.58 (0.59)
  Baseline to week 52 (n=226,223) | -8.92 (0.57) | -7.85 (0.57)

7. Secondary Outcome: Change From Baseline in Mean Sitting Pulse Pressure (msPP)
Description: Mean sitting pulse pressure for each patient and visit was calculated as the difference between the calculated values of mean sitting systolic blood pressure and mean sitting diastolic blood pressure.
Time Frame: baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n=226,222) | -13.13 (0.82) | -8.86 (0.82)
  Baseline to week 52 (n= 226, 223) | -15.02 (0.79) | -13.58 (0.80)

8. Secondary Outcome: Change From Baseline in Mean Arterial Pressure (MAP)
Description: Mean arterial pressure (MAP) was calculated from mean sitting systolic BP (msSBP) and mean sitting diastolic BP (msDBP) as (2 * msDBP + msSBP)/3.
Time Frame: baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n=226, 222) | -12.19 (0.68) | -8.57 (0.68)
  Baseline to week 52 (n=226, 223) | -13.92 (0.63) | -12.38 (0.64)

9. Secondary Outcome: Change From Baseline in Mean 24-hour Systolic Blood Pressure (maSBP)
Description: An Ambulatory Blood Pressure Monitor (ABPM) measured a participant's blood pressure over a 24 hour period using an automated validated monitoring device at baseline, week 12 and at week 52 starting one day before each visit. The 24 hour maSBP was calculated by taking the mean of all ambulatory systolic blood pressure readings for the 24 hour period.
Time Frame: Baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n= 164, 162) | -13.25 (0.62) | -9.14 (0.62)
  Baseline to week 52 (n= 174, 176) | -14.15 (0.59) | -14.32 (0.58)

10. Secondary Outcome: Change From Baseline in Mean 24-hour Diastolic Blood Pressure (maDBP)
Description: An Ambulatory Blood Pressure Monitor (ABPM) measured a participant's blood pressure over a 24 hour period using an automated validated monitoring device at baseline, week 12 and at week 52 starting one day before each visit. The 24 hour maDBP was calculated by taking the mean of all ambulatory systolic blood pressure readings for the 24 hour period.
Time Frame: Baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to week 12 (n= 164, 162) | -7.44 (0.37) | -5.48 (0.36)
  Baseline to week 52 (n= 174, 176) | -8.85 (0.35) | -8.44 (0.34)

11. Secondary Outcome: Change From Baseline in Mean 24-hour Ambulatory Pulse Pressure (maPP)
Description: Mean 24 hour ambulatory pulse pressure was calculated as the difference between the mean 24 hour systolic and diastolic ambulatory blood pressure in corresponding visits i.e. baseline, week 12 and week 52.
Time Frame: Baseline, 12 weeks, and 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Number analyzed (Participants) | 229 | 225
mmHg
  Baseline to Week 12 (n=164, 162 ) | -5.77 (0.35) | -3.69 (0.35)
  Baseline to week 52 (n=174, 176) | -5.26 (0.36) | -5.91 (0.35)

ADVERSE EVENTS:
Arm/Group | LCZ696 (Sacubitril/Valsartan) | Olmesartan
Serious Adverse Events (participants affected / at risk) | 16/229 | 13/225
Other Adverse Events (participants affected / at risk) | 73/229 | 55/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=229) | Olmesartan (N=225)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0
DOUGLAS' ABSCESS (Infections and infestations) | 1 | 0
PERITONITIS (Infections and infestations) | 1 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
PULMONARY CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BRAIN STEM INFARCTION (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY PNEUMATOCELE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (Sacubitril/Valsartan) (N=229) | Olmesartan (N=225)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 1
DIARRHOEA (Gastrointestinal disorders) | 6 | 5
NAUSEA (Gastrointestinal disorders) | 5 | 2
OEDEMA PERIPHERAL (General disorders) | 6 | 2
INFLUENZA (Infections and infestations) | 7 | 5
NASOPHARYNGITIS (Infections and infestations) | 16 | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 10
DIZZINESS (Nervous system disorders) | 12 | 12
HEADACHE (Nervous system disorders) | 14 | 10
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 2
HYPOTENSION (Vascular disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.